CLINICAL TRIAL: NCT04791254
Title: Anorexia iN Cancer Patients: Assessment of the Gut HORmone and Cytokine Profile and Body Composition, and the Impact of Dietetic Support in Patients With Gastrointestinal Cancer. (ANCHOR Study)
Brief Title: Anorexia iN Cancer Patients: ANCHOR
Acronym: ANCHOR
Status: Recruiting | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other); Manchester Metropolitan University (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp141
Record Dates: First submitted 2021-02-24; First posted 2021-03-10 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Gastric Cancer; Oesophageal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- A - main study cohort: This is the main study cohort. All patients with upper gastrointestinal (gastric, oesophageal and gastro-oesophageal) cancers attending the medical oncology clinic and commencing systemic therapy will be invited to participate.
  They will receive dietician support as part of their standard treatment. They will undergo assessments of body composition as part of this assessment
- Sub-cohort B: This sub-cohort will be invited to undergo more detailed fitness testing in the form of cardio-pulmonary exercise testing in addition to their routine care in the main cohort
- sub-cohort C: This sub-cohort will be invited to undergo an assessment of gut hormone and cytokine levels in addition to their routine care in the main cohort
- Cohort D: This is a cohort of healthy volunteers invited to act as a control to cohort C and undergo the gut hormone assessment

SUMMARY:
The rationale for this study is to prospectively investigate the outcomes of patients undergoing standard dietetic interventions alongside treatment for their advanced gastrointestinal cancers, and to further characterise the relationship with body composition.

A number of patients will be enrolled in a sub-study investigating the neuronal-enteroendocrine-hypothalamic axis.

Gut hormone study. Our hypothesis is that proinflammatory cytokines produced by the tumour can not only affect appetite directly through the vagal and the central melanocortin system but also indirectly though the enhanced EEC activity; either through increased number or increased function.

In this study, the investigators will explore and compare the pattern and levels (pre-prandial and post prandial) of the pro-inflammatory cytokines and gut hormones between stage-standardised anorexic and non-anorexic cancer patients and age-matched healthy controls.

DETAILED DESCRIPTION:
Poor nutritional status contributes significantly to poor outcomes in patients with upper GI cancers, in some patients, directly leading to death. Poor fitness, in terms of reduced muscle mass (sarcopenia) or physical performance, is associated with higher treatment toxicity and poor treatment outcomes.

However the relationship between different markers of nutritional status and body composition with fitness is not fully understood. It is also not known what impact dietetic interventions have on the reduced survival seen in patients with weight loss at baseline.

Finally, the underlying interaction between the neuronal-enteroendocrine-hypothalamic axis that regulates appetite is poorly understood but believed to be impaired in patients with upper GI cancers because of a number of altered mechanisms.

Therefore the rationale for this study is to prospectively investigate the outcomes of patients undergoing standard dietetic interventions alongside treatment for their advanced gastrointestinal cancers, and to further characterise the relationship with body composition.

A number of patients will be enrolled in a sub-study investigating the neuronal-enteroendocrine-hypothalamic axis.

The hypothesis is that proinflammatory cytokines produced by the tumour can not only affect appetite directly through the vagal and the central melanocortin system but also indirectly though the enhanced EEC activity; either through increased number or increased function.

In this study, the investigators will explore and compare the pattern and levels (pre-prandial and post prandial) of the pro-inflammatory cytokines and gut hormones between stage-standardised anorexic and non-anorexic cancer patients and age-matched healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: Cohort A

  1. Patients with stage IV gastric or GOJ adenocarcinoma or locally advanced non-resectable adenocarcinoma
  2. Histologically proven adenocarcinoma, squamous cell carcinoma or poorly differentiated carcinoma
  3. Patients should be chemotherapy or immune therapy naïve (for their current diagnosis).
  4. Patient must be 18 years of age or above.
  5. Patient must be able to understand the study information given to them and be willing to give consent for trial participation.
  6. Patients should be commencing a course of palliative chemotherapy treatment with the upper GI team at the Christie Hospital

In addition the above patients enrolled in cohort B must meet the following criteria

Inclusion criteria: Cohort B

1. Be physically able to perform moderate exercise (to their own tolerance) on a stationary bicycle or treadmill

In addition to the above patients in cohort C must meet the following criteria

Inclusion Criteria: Cohort C

1. Histologically proven adenocarcinoma or poorly differentiated carcinoma
2. Patients should be chemotherapy or immune therapy naïve.
3. Patients must be able and willing to fast for 8-10 hours. 4 5.1 Patients in the anorexic group must have completed the FAACT AC/S questionnaire and scored ≤24 in total score and ≤ 2 in the appetite specific question.

5.2 For inclusion in the non-anorexic group patients must have completed the FAACT AC/S questionnaire; the total score should be > 37 and ≥3 for the appetite specific question.

Inclusion criteria: Cohort D - healthy controls

1. Participants must be 18 years of age or above.
2. Participants must be able and willing to fast for 8-10 hours.
3. Participants must be able to understand the study information given to them and be willing to give consent for trial participation.
4. Participants must have completed the FAACT AC/S questionnaire and scored ≤24 in total score and ≤ 2 in the appetite specific question, for the anorexic group. For inclusion in the non-anorexic group the total score should be > 37 and ≥3 for the appetite specific question.

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:

Exclusion criteria Cohort A:

1. Patients unable to give informed consent
2. Patients not undergoing systemic anti-cancer treatment at The Christie hospital, for example patients not deemed fit enough for treatment, patients having alternative treatments such as radiotherapy or surgery, or patients referred for 2nd opinions.

Exclusion criteria Cohort B:

1. Recent myocardial infarction or stroke
2. Recent abdominal, eye or thoracic surgery
3. A recent respiratory tract infection (within 3 weeks)
4. Any chest pain on the day of the test
5. A positive COVID-19 test

Exclusion Criteria Cohort C & D : all patients and healthy volunteers

1. Symptoms of dysphagia of any cause, oesophageal or gastric obstruction (assessed via medical history/O'Rourke score). Patients with O'Rourke score ≥2 will be excluded.
2. Presence of oesophageal stent or any other kind of feeding aid (nasogastric tube, nasoduodenal tube, gastrostomy, jejunostomy)
3. Presence of brain metastases or any kind of brain tumor including benign pituitary adenomas.
4. Histological diagnosis of neuroendocrine tumor, or mixed tumor.
5. Previous gastro-duodenal surgery.
6. History of Inflammatory Bowel Disease (Ulcerative colitis, Crohn's disease).
7. History of Coeliac disease.
8. History of endocrine disease (Diabetes mellitus, Thyroid disease, Cushing's)
9. Significant past or present eating disorder e.g. anorexia nervosa, bulimia nervosa.
10. Current active infection (general or intestinal).
11. Chronic use of immunomodulatory drugs (steroids, immunosuppressant drugs, recent use of corticosteroids would require a two week washout period prior to study assessments).
12. Chronic use of NSAIDS or aspirin. (Periodic use can be accepted).
13. Patients with pacemakers. (Contraindication for BIA).
14. Allergy to any of the ingredients of the meal test or unwillingness to consume the particular meal (Heinz Chicken soup or Heinz Mushroom soup).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with advanced (either metastatic, or locally advanced and inoperable) gastro-oesophgeal (including primary oesophageal, gastro-oesophageal junction or gastric) cancer, presenting to undergo first line systemic therapy
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Survival outcomes in patients with advanced upper gastrointestinal cancers receiving dietetic interventions. | Through study completion, median expected overall survival < 1 year.
  Progression free and overall survival from diagnosis.
Differences in patterns of plasma gut hormone and cytokine levels as measured by ELISA between study participants. | 3 months from completion of data collection
  Plasma gut hormones and cytokine levels as measured via ELISA including, ghrelin, insulin, GLP-1, PYY, pancreatic polypeptide, GIP, CHromogranin A, CCK. The following cytokines will be included. IL-1, IL-6, TNF-α

SECONDARY OUTCOMES:
Correlation between hormonal and cytokine profile and body composition as measured by bioelectrical impedance analysis and CT measured muscle mass (for patients only) and density. | Within 6 months of completion of data collection
Correlation between nutritional status, body composition and physical fitness | Within 6 months of completion of data collection

CONTACTS AND LOCATIONS:
Overall Officials: Was Mansoor, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No